CLINICAL TRIAL: NCT04360616
Title: The Diagnosis and Prognosis of Nonpalpable Breast Cancer Detected by the Ultrasound vs Mammography: a Clinical Noninferiority Trial.
Brief Title: The Diagnosis and Prognosis of Nonpalpable Breast Cancer Detected by the US vs Mammography: a Clinical Noninferiority Trial.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of the Fourth Military Medical University (Other)
Responsible Party: Principal Investigator, Song Hongping, Principal Investigator, The First Affiliated Hospital of the Fourth Military Medical University
Other Study IDs: US-MAM
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- MG+: the lesion could detected by mammography
  Interventions: Diagnostic Test: imaging
- US+: the lesion could detected by breast ulrtasound
  Interventions: Diagnostic Test: imaging

INTERVENTIONS:
Diagnostic Test: imaging — perform US and mammography examination

SUMMARY:
To evaluate and compare the sensitivity, specificity, AUC, pathology results of core needle biopsy and surgical pathology results coincidence rate, tumor staging, and DFS (disease-free survival) of US-detected nonpalpable breast cancer vs mammography-detected nonpalpable breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 years and over with full capacity for civil conduct;
2. Breast imaging examination (including mammography and breast ultrasound) found that patients with BI-RADS 4 or nonpalpable lesion need to have breast biopsy (refer to the classification of BI-RADS, which is consistent with the indications for biopsy), including some patients with BI-RADS 3 nonpalpable breast lesions who are willing to have biopsy;
3. Voluntarily participate in and sign the informed consent form, and be willing to accept the inspection designated by this test;
4. The results of blood examination, coagulation examination, preoperative infection examination, and 12 lead ECG examination within 2 weeks before biopsy met the biopsy requirements;
5. It conforms to the biopsy standard (refer to the image-guided breast histology biopsy guide in the breast cancer diagnosis and treatment guide and specification of China Anti Cancer Association (2019 version)).

Exclusion Criteria:

1. Women are participating in another clinical trial of drug or medical device;
2. Women with neuropsychiatric disorders;
3. Women with severe systemic diseases and serious bleeding diseases that can not cooperate with the examination, or the researchers think it is not suitable to participate in this clinical trial;
4. Other subjects not suitable for X-ray examination

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Female patients over 18 years old from China
Sampling Method: Probability Sample
Enrollment: 1277 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Sensitive | 3 days
  Proportion of corrected-detected malignant lesions by the US or MG
Specificity | 3 days
  Proportion of corrected-detected benign lesions by the US or MG
Area under curve | 3 days
  Area under receiver operating characteristic (ROC) curve in percentage (%)
Disease-free survival (DFS) | 3 years
  The time that the patient is free of the signs and symptoms of a disease after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hongping Song, MD, Principal Investigator — Xijing hospital of The fourth military medical university
Locations (1):
- The First Affiliated Hospital of Fourth Military Medical University, Xi'an, Shaanxi, China